CLINICAL TRIAL: NCT06828926
Title: Project Gnosis: the Neural, Physical, and Psychosocial Processes and Health Outcomes of an 8-week Tai Chi Intervention in Older Adults with and Without Mild Cognitive Impairment
Brief Title: Project Gnosis: the Neurophysical and Psychosocial Health Outcomes of Tai Chi for Older Adults with Cognitive Concerns or Mild Cognitive Impairment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Ohio_U_FY25-124
Record Dates: First submitted 2025-01-13; First posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-02

CONDITIONS: Mild Cognitive Impairment (MCI); Sarcopenia
Keywords: Tai Chi; Cognitive Function
MeSH Terms: conditions — Cognitive Dysfunction; Sarcopenia | interventions — Tai Ji

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Tai Chi (Experimental): The Tai Chi program content is based on the Harvard Medical School (HMS) Guide to Tai Chi, developed by clinical scientist Dr. Peter M. Wayne. Each participant will receive a workbook that describes the philosophy, evidence, and practice of Tai Chi, along with a video series for home practice that features the exercises from the HMS Guide to Tai Chi program. The in-person classes will be led by the Principal Investigator (PI) and delivered weekly over 8 weeks, with 75-minute sessions. The in-person and video series will introduce practice principles and tips on establishing and maintaining a practice, followed by a series of warm-up exercises, Tai Chi movements, and cool-down exercises.
  Interventions: Behavioral: Tai Chi

INTERVENTIONS:
Behavioral: Tai Chi — The Tai Chi program content is based on the Harvard Medical School (HMS) Guide to Tai Chi, developed by clinical scientist Dr. Peter M. Wayne. Each participant will receive a workbook that describes the philosophy, evidence, and practice of Tai Chi, along with a video series for home practice that features the exercises from the HMS Guide to Tai Chi program. The in-person classes will be led by the PI and delivered weekly over 8 weeks, with 75-minute sessions. The in-person and video series will include an introduction to the principles of practice and tips on establishing and maintaining a practice, followed by a series of warm-up exercises, Tai Chi movements, and cool-down exercises. The Tin-person (and offer virtual live sessions for those who cannot attend in-person) over 8 weeks, accompanied by a workbook and video-recorded practices to promote self-management.

SUMMARY:
Mild Cognitive Impairment (MCI) in older adults is linked to muscle loss (sarcopenia) and can lead to dementia, with pain further impacting cognitive and physical performance. Tai Chi, a mind-body exercise, is recommended for managing MCI as it supports cognitive function, mood, and physical health.

The investigators' first goal is to characterize the correlation of heart rate variability and cortical activity on cognitive function and the psychosocial correlates of pain interference and social isolation on cognitive function at baseline and post-intervention (8 weeks of Tai Chi). The second goal is to explain the role of sarcopenia and obesity in the relationship between pain interference and cognitive function. The investigators also want to examine the index of the predictive capacity regarding sarcopenia and obesity on cognitive function outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Participants who are older adults, defined as ≥60 years old.
2. Participants must have the ability to independently stand without the use of an assistive device for 20 minutes.
3. People with Mild Cognitive Impairment (MCI) (initial cohort) and without MCI (age-gender matched healthy controls). A score of between >18 and ≤26 on the Montreal Cognitive Assessment (MoCA) will be used to classify MCI. A score above 26 is considered normal.

Exclusion Criteria:

1. Participants with significant uncontrolled medication, and cardiovascular, respiratory, and metabolic symptoms will be excluded from participation in the study, as these symptoms could impact their engagement with the engagement of Tai Chi.
2. Investigators will administer a brief screening questionnaire to assess (a) hypotension symptoms related to intensive treatment of hypertension and (b) hypoglycemia related to intensive treatment of diabetes, as these conditions are associated with cognitive decline.
3. Investigators will capture data on potential sleep apnea and administer the Stop-Bang Questionnaire to identify potential sleep-disordered breathing. Participants with significant uncontrolled sleep apnea will be excluded as this could also impact their engagement in the intervention and influence the primary outcome measure of cognitive function.

2. Currently or recently practicing Tai Chi. Participants will be excluded if they are currently practicing Tai Chi. If participants have previously engaged in Tai Chi, there will be a washout period of at least 6 months before considering enrollment in the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-12 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Executive Function - Stroop Color-Word Interference Test | From enrollment to the end of treatment at 8 weeks
  Delis-Kaplan Executive Function System Stroop Color-Word Interference Test
Executive Function - Semantic Fluency Test | From enrollment to the end of treatment at 8 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status - Semantic Fluency Test

SECONDARY OUTCOMES:
Cognitive Function - Processing Speed | From enrollment to the end of treatment at 8 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status Coding Test
Pain Interference | From enrollment to the end of treatment at 8 weeks
  Patient Reported Outcome Measurement Information System (PROMIS) - Pain Interference Item Bank
Social Isolation | From enrollment to the end of treatment at 8 weeks
  Patient Reported Outcome Measurement Information System (PROMIS) Social Isolation Item Bank
Positive Affect | From enrollment to the end of treatment at 8 weeks
  Patient Reported Outcome Measurement Information System (PROMIS) Positive Affect Item Bank
Meaning and Purpose | From enrollment to the end of treatment at 8 weeks
  Patient Reported Outcome Measurement Information System (PROMIS) Meaning and Purpose Item bank
Heart Rate Variability | From enrollment to the end of treatment at 8 weeks
  Heart Rate Variability recorded while sitting for 5 minutes using a photoplethysmogram.
Cortical activity | From enrollment to the end of treatment at 8 weeks
  Cortical activity will be recorded during a brief Tai Chi Practice before and after the 8-week Tai Chi intervention using a functional Near Infrared Spectroscopy system.

OTHER OUTCOMES:
Cognitive Assessment Screen | From enrollment only
  Montreal Cognitive Assessment used as a screening tool which measures short term memory, visuospatial abilities, executive functions, attention, concentration and working memory, and language orientation to time and place.
Body Mass Index | From enrollment only
  Body Mass Index (BMI) will be assessed to identify the moderating role of obesity on pain interference and executive function. Weight and height will be combined to report BMI in kg/m^2).
Physical Performance Test Battery for Sarcopenia (1 of 6) | From enrollment to the end of treatment at 8 weeks
  (1) Hand Grip Strength using a JAMAR® dynamometer, adjusted to fit participants' hands as described elsewhere. A minimum of three trials with 60 seconds of rest between trials, and additional trials if the highest two values differ by more than 3 kg. Unit: Force in kilograms
  The investigators will diagnose sarcopenia using the European Working Group's (EWGSOP2) revised consensus definition, which involves assessing two measures and current sarcopenia reference values: (i) hand grip strength via dynamometry and (ii) gait speed.
Physical Performance Test Battery for Sarcopenia (2 of 6) | From enrollment to the end of treatment at 8 weeks
  (2) Usual Gait Speed over 4 meters to assess for gait speed. Unit: Seconds
  The investigators will diagnose sarcopenia using the European Working Group's (EWGSOP2) revised consensus definition, which involves assessing two measures and current sarcopenia reference values: (i) hand grip strength via dynamometry and (ii) gait speed.
Physical Performance Test Battery for Sarcopenia (3 of 6) | From enrollment to the end of treatment at 8 weeks
  (3) Six Minute Walk Test to assess for submaximal aerobic walking capacity. Unit: Meters
Physical Performance Test Battery for Sarcopenia (4 of 6) | From enrollment to the end of treatment at 8 weeks
  (4) Four-Square Step Test to assess for dynamic balance that involves stepping over objects forward, sideways, and backward. Unit: Seconds
Physical Performance Test Battery for Sarcopenia (5 of 6) | From enrollment to the end of treatment at 8 weeks
  (5) 5x Repeated Sit-to-Stand Test to assess lower extremity strength. Unit: Seconds
Physical Performance Test Battery for Sarcopenia (6 of 6) | From enrollment to the end of treatment at 8 weeks
  (6) Stair Climb Power Test to assess lower extremity power. Unit: Seconds.

CONTACTS AND LOCATIONS:
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
There is a plan to make individual participant data (IPD) collected in this study, including data dictionaries, available to other researchers after the end of the study after de-identification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.